CLINICAL TRIAL: NCT04045418
Title: A Study on the Microcirculatory Characteristics of Meridian Phenomenon for the Heart and Lung Meridians Based on Patients With Chronic Obstructive Pulmonary Disease
Brief Title: A Study on the Microcirculatory Characteristics of Meridian Phenomenon for the Heart and Lung Meridians Based on Patients With COPD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhejiang Chinese Medical University (Other Government)
Collaborators: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other); The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Jianqiao Fang, President, Zhejiang Chinese Medical University
Other Study IDs: 2019ZY004-MERIDIAN
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: meridians; acupuncture; chronic stable angina pectoris; meridian phenomenon; laser doppler
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Laser-Doppler Flowmetry; Moxibustion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COPD group: This group will include 40 patients with chronic obstructive pulmonary disease (COPD).
  Interventions: Device: Laser doppler
- Healthy control group: This group will include 40 healthy volunteers.
  Interventions: Device: Laser doppler
- Healthy intervention group: This group will include 40 healthy volunteers. Two sessions of moxibustion intervention will be performed in the Heart meridian and Lung meridian successively. The washout period between the two sessions is at least one day.
  Interventions: Device: Laser doppler

INTERVENTIONS:
Device: Laser doppler — A laser doppler flowmetry will be used to measure the microcirculatory characteristics of meridian phenomena. The probes will be left at relevant measuring sites. Blood flow curve and Perfusion units (PU ) will be recorded constantly.
  1. Healthy control group and COPD group The probes will be left at Shenmen (HT7) and Shaohai (HT3) of the Heart meridian, Taiyuan (LU9) and Chize (LU5) of the Lung meridian for 5 minutes.
  2. Healthy intervention group Two sessions of moxibustion will be performed in the Heart meridian and Lung meridian successively.
  Other Names: moxibustion

SUMMARY:
Although some important progresses were made in the field of the meridian research, no breakthroughs have been achieved. Besides,there are some problems in meridian researches. Particularly, previous research of meridian phenomenon involved lots of subjective elements and outcomes.Researches that use modern scientific techniques to investigate the biological characteristics of meridian phenomenon are urgently needed. Therefore, this study is designed to assess the microcirculatory characteristics of meridian phenomenon for the Heart and Lung meridians by using laser doppler. Thus, the biological characteristics of meridian phenomenon could be presented objectively in a scientific methodology

DETAILED DESCRIPTION:
This study will include 40 patients diagnosed with chronic obstructive pulmonary disease (COPD) and 80 healthy volunteers. Laser doppler examination will be adopted to assess the microcirculatory characteristics of meridian phenomenon for Heart and Lung meridians in the physiology/pathological state. Moreover, the site specificity for the meridian-visceral association and surface-surface association between the Heart and Lung meridians will be investigated.Primary outcomes will be blood flow curve and blood perfusion units(PU).Furthermore, this study will build standardized techniques and schemes for detecting the microcirculatory characteristics of meridian phenomenon for Heart and Lung meridians. The results of this study could also provide scientific foundation for traditional meridian theories.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the COPD group

1. Patients should meet the above diagnostic criteria, and the severity of COPD is in the stage of GOLD 2 or 3 based on pulmonary function testing;
2. COPD patients in the stable phase, who present with mild symptoms of cough, expectoration and short breath;
3. 35 ≤ age ≤75 years, male or female;
4. Patients have clear consciousness and could communicate with others normally;
5. Patients could understand the full study protocol and have high adherence.Written informed consent is signed by themselves or their lineal kin.

Inclusion criteria for health volunteers

1. Healthy volunteers who could provide a recent (in the past 3 month) medical examination report to confirm they have not any cardiovascular, respiratory, digestive, urinary, hematological, endocrine and neurological disease;
2. age ≥20 years, male or female;
3. Participants have clear consciousness and could communicate with others normally;
4. Participants could understand the full study protocol and have high adherence .Written informed consent is signed by themselves or their lineal kin.

Exclusion Criteria:

Exclusion criteria for the COPD group

1. Patients who fail to meet the diagnostic criteria for COPD, or COPD patients in the phase of acute exacerbation;
2. Patients have the following complications, which includes pneumonia, bronchial asthma, bronchiectasis, active tuberculosis, pneumothorax, chest trauma, tumors of the lung or thorax, and other confirmed respiratory diseases;
3. Patients have concomitant conditions of heart diseases, such as chronic stable angina pectoris (CSAP);
4. Patients have serious concomitant conditions and fail to treat them effectively, such as diseases of the digestive, urinary, respiratory, hematological, and nervous system;
5. Patients have mental illness, severe depression, alcohol dependence or history of drug abuse;
6. Pregnant or lactating patients; Patients are participating in other trials.

Exclusion criteria of health volunteers

1. Participants have sudden severe diseases during the trial, such as cardiovascular diseases, liver diseases, kidney diseases, urinary diseases and hematological diseases.
2. Participants have mental illness, severe depression, alcohol dependence or history of drug abuse;
3. Pregnant or lactating participants ;
4. Participants are participating in other trials.

Ages: 20 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 40 patients with chronic obstructive pulmonary disease (COPD)and 80 healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Blood flow curve | 5 minutes of baseline, 15 minutes during moxibustion and 5 minutes after stopping moxibustion.
  The blood flow curve could reflect the microcirculatory flux in the measuring sites.
Blood perfusion units | 5 minutes of baseline, 15 minutes during moxibustion and 5 minutes after stopping moxibustion.
  Perfusion units (PU)=concentration of moving blood cells (CMBC)×velocity (V)

CONTACTS AND LOCATIONS:
Overall Officials: Jianqiao Fang, Principal Investigator — Zhejiang Chinese Medical University
Locations (1):
- the Third affiliated hospital of Zhejiang Chinese Medical university, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hsiu H, Huang SM, Chao PT, Jan MY, Hsu TL, Wang WK, Wang YY. Microcirculatory characteristics of acupuncture points obtained by laser Doppler flowmetry. Physiol Meas. 2007 Oct;28(10):N77-86. doi: 10.1088/0967-3334/28/10/N01. Epub 2007 Sep 18. PMID 17906382
- [Background] Hsiu H, Hsu WC, Chen BH, Hsu CL. Differences in the microcirculatory effects of local skin surface contact pressure stimulation between acupoints and nonacupoints: possible relevance to acupressure. Physiol Meas. 2010 Jun;31(6):829-41. doi: 10.1088/0967-3334/31/6/007. Epub 2010 May 18. PMID 20479520
- [Background] Hsiu H, Hsu WC, Hsu CL, Huang SM, Jan MY, Wang WK, Wang YY. Spectral analysis on the microcirculatory laser Doppler signal at the acupuncture point. Annu Int Conf IEEE Eng Med Biol Soc. 2008;2008:1084-6. doi: 10.1109/IEMBS.2008.4649348. PMID 19162851
- [Background] Hsiu H, Hsu WC, Hsu CL, Huang SM, Lin YY. Microcirculatory changes by laser Doppler after infrared heating over acupuncture points--relevance to moxibustion. Photomed Laser Surg. 2009 Dec;27(6):855-61. doi: 10.1089/pho.2008.2390. PMID 19698003
- [Background] Hsiu H, Huang SM, Chao PT, Hsu WC, Hsu CL, Jan MY, Wang WK, Wang YY. Study on the microcirculatory blood velocity of acupoint monitored by laser Doppler signal. Annu Int Conf IEEE Eng Med Biol Soc. 2007;2007:959-62. doi: 10.1109/IEMBS.2007.4352451. PMID 18002117
- [Background] Litscher G, Wang L, Huber E, Nilsson G. Changed skin blood perfusion in the fingertip following acupuncture needle introduction as evaluated by laser Doppler perfusion imaging. Lasers Med Sci. 2002;17(1):19-25. doi: 10.1007/s10103-002-8262-9. PMID 11845364
- [Background] Hsiu H, Hsu WC, Huang SM, Hsu CL, Lin Wang YY. Spectral analysis of the microcirculatory laser Doppler signal at the Hoku acupuncture point. Lasers Med Sci. 2009 May;24(3):353-8. doi: 10.1007/s10103-008-0569-8. Epub 2008 May 27. PMID 18504639
- [Background] Huang T, Wang RH, Zhang WB, Han B, Wang GJ, Tian YY, Zhang YQ. The influence of different methods of acupuncture on skin surface perfusion. J Tradit Chin Med. 2012 Mar;32(1):40-4. doi: 10.1016/s0254-6272(12)60029-6. PMID 22594100

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/18/NCT04045418/Prot_SAP_002.pdf
  • Informed Consent Form (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/18/NCT04045418/ICF_003.pdf